CLINICAL TRIAL: NCT03338985
Title: Role of Senescence in the Development of Endometrial Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PA17002
Record Dates: First submitted 2017-11-08; First posted 2017-11-09 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Endometrial Hyperplasia and Endometrial Cancers
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group "cases patients" (Experimental): patients with endometrial hyperplasia or endometrial cancers
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — Genetic analysis of the samples taken during the surgery (hysterectomy or curettage resection) using CGH array technique.

SUMMARY:
Several molecular studies showed chromosomal alterations in patients with endometrial cancer, with gains in 1q, 19p, 19q, 8q, 10q and 10p and loss of 4q, 16q and 18q. Several genes of interest have been identified (P53, PTEN, PIK3CA, ß-catenin, K-ras ...).

A study has already been carried out at the Reims University Hospital with inclusion of patients with endometrial cancer and patients with endometrial hyperplasia. It identified specific alterations of nosologic continuum of pathology and characterize areas of interest on the genome.

DETAILED DESCRIPTION:
make a pangenomic investigation of genetic abnormalities in atypical endometrial hyperplasia and endometrial cancers.

ELIGIBILITY:
Inclusion Criteria:

* patient with endometrial hyperplasia or endometrial cancer
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

- patient with neoadjuvant chemotherapy or radiotherapy prior to surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-10-16 (Estimated); Study Completion 2020-04-16 (Estimated)

PRIMARY OUTCOMES:
Genetic imbalances | Day 0
  Genetic aberrations detected by comparative genomic hybridization (CGH arry)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France